CLINICAL TRIAL: NCT01711203
Title: The Addition of a Pilates Program for Short-Term Improvements in Self Report and Physical Functions With Patients With Spondylolysis or Spondylolisthesis: A Randomized Clinical Trial
Brief Title: The Addition of a Pilates Program for Short-Term Improvements in Patients With Spondylolysis or Spondylolisthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Megan Donaldson PT, PhD, FAAOMPT (Other)
Collaborators: Akron Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Megan Donaldson PT, PhD, FAAOMPT, Assistant Professor, Walsh University
Organization: Walsh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Spondy 12-35
Record Dates: First submitted 2012-10-09; First posted 2012-10-22 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Spondylolisthesis; Spondylolysis; Children
Keywords: Spondylolysis; Spondylolisthesis; Rehabilitation; Physical Therapy; Children
MeSH Terms: conditions — Spondylolisthesis; Spondylolysis | interventions — Functional Laterality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motor Control (Experimental): Pilates-based exercise with verbal cues to facilitate motor control Plank progression, use of feedback tool VERBAL CUES FOR MOTOR CONTROL GROUP (could also include above cues) "Maintain neutral spine" "Not too arched, not too flexed" "Remember your pilates position" "Inhale, exhale" "Let me hear your breath"
  Interventions: Other: Motor Control
- General strengthening (Active Comparator): Patient group that will receive active strengthening without specific verbal cueing to recruit deeper abdominal musculature. Core strengthening and lower quarter strengthening is the focus of this group.
  Verbal cuing will include:
  VERBAL CUEING FOR NON-MOTOR CONTROL GROUP
  "Keep your back straight" "Don't slouch" "Don't arch your back" "Don't let your body move" "Nothing should move but your arms" "tighten up your abs" "suck in your stomach" "feet shoulder-width apart, knees bent, shoulders back, hold your stomach tight" Time will be kept the same as the intervention group.
  Interventions: Other: General Strengthening

INTERVENTIONS:
Other: Motor Control — Exercises and verbal cues to facilitate deep abdominal control and contraction for muscular stabilization/re-training.
  Arms: Motor Control
Other: General Strengthening — General abdominal and lower quarter musculature strengthening
  Arms: General strengthening

SUMMARY:
Purpose: To determine the effectiveness of an augmented Pilates program, when combined to a multimodal strengthening program, for patients under the age of 21, who have spondylolysis and/or spondylolisthesis.

Significance of the topic: Spondylolysis and spondylolisthesis are often diagnosed in children and adolescents presenting with low back pain.

A randomized, clinical trial, test-retest design, with a 3 week and 6 week assessment with functional performance test measures, exercise logs, adherence scale for patient and parent perception, and outcome measures (Global rating of change (GROC) and Modified Oswestry Disability Index (ODI)). This study will attempt to obtain at least 120 subjects that will be randomized into two groups: bracing and a general strengthening program vs. bracing and a Pilates/motor learning program combined with a general strengthening program.

This study will begin with an initial examination and continue with treatment sessions 2x/week for 6 weeks. A follow up phone call will be conducted at 3 months after completing the 6-week protocol. The follow up phone call will be an oral conducted GROC and ODI outcome measures.

DETAILED DESCRIPTION:
Location: Akron Children's Hospital, Sports Medicine. For research purposes, the study will conclude at the end of the 6 weeks, however, if the patient has not met their physical therapy goals, then physical therapy may continue upon collaboration with the patient and his/her parents (if a minor), physical therapist, and referring physician.

Initially, there will be a letter to discuss the opportunity to participate in the research study within initial intake paperwork. This will allow the patient and parent to have some preliminary information prior to consulting with the therapist. As is customary, the patient will be assigned to a licensed PT for the initial examination. The initial examining therapist will be responsible to discuss and provide the patient with the pre-enrollment information and informed consent (estimation of time needed approximately 15 minutes) and may obtain consent any time after the pre-enrollment discussion or until the start of the patient's second session. Upon agreement of participation in the study, the patient will be able to complete the additional paperwork required as part of the study (outcome measures). The patient will be randomized after self-inclusion in to the study into one of two groups by role of dice where 1, 3, 5 is the intervention group and 2, 4, 6 is the clinical control group.

The initial examination will include a subjective history taking, and objective assessment with physical testing of the spine including active range of motion, passive range of motion, strength assessment/endurance assessment of the lumbar musculature. The examination will take approximately 45 minutes to 1 hour in length.

Description of Subjects (include age range, selection criteria, recruitment procedures, anticipated and desired sample size)-

Subjects of the ages 8-21 are eligible to participate in this study. Due to the inclusion of a vulnerable subject the responsible party/parent or guardian must grant inclusion and must be able to attend the initial physical therapy evaluation of the minor and sign all consenting documents. The physician offices within the surrounding hospital area and doctors that typically refer to this clinic will be notified of the research study (attachment physician letter and flyer for the facility). Patients will be included in the study if they meet the following criteria:

1. Age of subject must be between 8-21 years old
2. Ability to read and understand the English language
3. Parent/caregiver consent
4. Written medical diagnosis of spondylolysis or spondylolithesis from the physician with or without imaging.

The investigators plan to target a maximum of 120 subjects for the large study, allowing a 20% drop out rate. This study is powered at n=100 subjects for at least a minimal effect to be calculated.

The investigators hypothesize a minimal effect on the patient group who receives the investigational "motor control" or Pilates based exercise compared to the general core strengthening program patient group.

Outcome Measures:

Numeric Pain Rating Scale

The numeric pain rating scale (NPRS) was used to capture the patient's level of pain. Patients were asked to indicate the intensity of current, best, and worst levels of pain over the past 24 hours using an 11-point scale ranging from 0 ("no pain") to 10 ("worst pain imaginable"). The average of the three ratings was used to represent the patient's level of pain over the previous 24 hours. This procedure has been shown to have adequate reliability, validity, and responsiveness in patients with LBP and has a minimally clinical important difference of 2-point change in patients with mechanical low back pain.

Global Rating of Change Scale

At the follow-up evaluation, each patient will complete a global rating of change (GROC). Patients will rate their overall perception of improvement since beginning treatment on a scale ranging from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). It has been recommended that scores on the GROC between ±3 and ±1 represent small changes; scores between ±4 and ±5 represent moderate changes, and scores of ±6 or ±7 large changes.

The Modified Oswestry Disability Questionnaire (ODI)

The Modified ODI is a self-administered questionnaire that requires 5 minutes to complete and 1 minute to score. Scores are associated with degree of disability ranging from minimal to bedbound. The ODI is a condition-specific disability scale for patients with LBP, consisting of 10 items addressing different aspects of function, each scored from 0-5 with higher values representing greater disability. This modified ODI has been found to have high levels of reliability, validity, and responsiveness. The MCID for the ODI has been identified at six points .On this scale, 0-20 equates to minimal disability, 20-40 moderate disability, 40-60 severe disability, 60-80 crippled, and 80-100 bed-bound or exaggerating.

Physical Endurance Tests/Measures McGill has established a performance test to examine the endurance profiles of healthy young men and women for the spine stabilizing musculature. Given the growing support for quantification of endurance, these data of endurance times and their ratios between extensor, flexor, and lateral flexor groups in healthy normal subjects are useful for patient evaluation and for providing clinical training targets. To establish isometric endurance holding times, as well as ratios between torso extensors, flexors, and lateral flexors (stabilizers), for clinical assessment and rehabilitation targets. The tests proved reliable, with reliability coefficients of >.97 for the repeated tests on 5 consecutive days and again 8 weeks later.

ELIGIBILITY:
Inclusion Criteria:

1. Age of subject must be between 8-21 years old
2. Ability to read and understand the English language
3. Parent/caregiver attendance and consent for initial evaluation
4. Written medical diagnosis of spondylolysis or spondylolithesis from the physician with or without imaging

Exclusion Criteria:

1. Not meeting the inclusion criteria
2. Not able to attend therapy 2x's per week
3. If physician prescription requests only physical bracing as rendered treatment
4. If patient presents with signs of neurological compromise
5. Red flags during the medical screening that would require the patient to see the physician

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Global Rating of Change Scale | 3 and 6 weeks and 3 months post discharge
  Patients will rate their overall perception of improvement since beginning treatment on a scale ranging from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). It has been recommended that scores on the GROC between ±3 and ±1 represent small changes; scores between ±4 and ±5 represent moderate changes, and scores of ±6 or ±7 large changes .

SECONDARY OUTCOMES:
Modified Oswestry Disability Index | Initial evaluation, 3 and 6 weeks and 3 months post discharge
  The Modified ODI is a self-administered questionnaire that requires 5 minutes to complete and 1 minute to score. Scores are associated with degree of disability ranging from minimal to bedbound. The ODI is a condition-specific disability scale for patients with LBP, consisting of 10 items addressing different aspects of function, each scored from 0-5 with higher values representing greater disability. This modified ODI has been found to have high levels of reliability, validity, and responsiveness . The MCID for the ODI has been identified at six points .On this scale, 0-20 equates to minimal disability, 20-40 moderate disability, 40-60 severe disability, 60-80 crippled, and 80-100 bed-bound or exaggerating.

OTHER OUTCOMES:
McGill's Physical Endurance Test Cluster | Initial evaluation, 3 weeks and 6 weeks
  McGill has established a performance test to examine the endurance profiles of healthy young men and women for the spine stabilizing musculature . Given the growing support for quantification of endurance, these data of endurance times and their ratios between extensor, flexor, and lateral flexor groups in healthy normal subjects are useful for patient evaluation and for providing clinical training targets. To establish isometric endurance holding times, as well as ratios between torso extensors, flexors, and lateral flexors (stabilizers), for clinical assessment and rehabilitation targets. The tests proved reliable, with reliability coefficients of >.97 for the repeated tests on 5 consecutive days and again 8 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Megan B Donaldson, PT PhD, Principal Investigator — Walsh University
Locations (1):
- Akron Children's Hospital Orthopaedic and Sports Physical Therapy Center, Akron, Ohio, United States

REFERENCES:
- [Background] Dreisinger TE, Nelson B. Management of back pain in athletes. Sports Med. 1996 Apr;21(4):313-20. doi: 10.2165/00007256-199621040-00006. PMID 8726348
- [Background] Klein G, Mehlman CT, McCarty M. Nonoperative treatment of spondylolysis and grade I spondylolisthesis in children and young adults: a meta-analysis of observational studies. J Pediatr Orthop. 2009 Mar;29(2):146-56. doi: 10.1097/BPO.0b013e3181977fc5. PMID 19352240
- [Background] Cavalier R, Herman MJ, Cheung EV, Pizzutillo PD. Spondylolysis and spondylolisthesis in children and adolescents: I. Diagnosis, natural history, and nonsurgical management. J Am Acad Orthop Surg. 2006 Jul;14(7):417-24. doi: 10.5435/00124635-200607000-00004. PMID 16822889